CLINICAL TRIAL: NCT03287570
Title: Clinical Research on the Efficacy and Safety of Cettum on Knee Osteoarthritis
Brief Title: Efficacy and Safety of Cettum for Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Eun Jung Kim (Other)
Collaborators: DongGuk University (Other)
Responsible Party: Sponsor-Investigator, Eun Jung Kim, Principle Investigator, DongGuk University
Organization: DongGuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DUBH2017-0002
Record Dates: First submitted 2017-09-13; First posted 2017-09-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; Moxibustion
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cettum (Electric moxibustion) (Experimental): The patients in this group receive Cettum (Electric moxibustion) treatment prescribed by a certified Korean Medicine Doctor with more than 6 years of Oriental Medicine College education.
  Interventions: Device: Cettum
- Traditional indirect moxibustion (Active Comparator): The patients in this group receive traditional indirect moxibustion treatment using the same points, applied by a certified Korean Medicine Doctor with more than 6 years of Oriental Medicine College education.
  Interventions: Procedure: Traditional indirect moxibustion
- Usual care (Other): The patients in this group maintain the usual treatment and self-care.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Cettum — The treatment is applied twice a week for 15 minutes for 6 weeks (12 sessions). 6 points (ST36, ST35, EX-LE4, SP9, SP10, ST34) are used for all the patients assigned to this group and investigator can be added up to 2 points depending on the patient condition. Electric moxibustion, Cettum (20X28X18mm) manufactured by K-medical Co.(Korea) is used.
  Other Names: Electric moxibustion
  Arms: Cettum (Electric moxibustion)
Procedure: Traditional indirect moxibustion — The treatment is applied twice a week for 6 weeks (12 sessions). 6 points (ST36, ST35, EX-LE4, SP9, SP10, ST34) are used for all the patients assigned to this group and investigator can be added up to 2 points depending on the patient condition. Traditional indirect moxibustion, Taekeukttum manufactured by Haenglim Seowon Medical Co.(China) is used. A total of three moxibustion cones are applied indirectly to each point per treatment session.
  Arms: Traditional indirect moxibustion
Other: Usual care — The patients in this group maintain the usual treatment and self-care.
  Arms: Usual care

SUMMARY:
The purpose of this study is verify the efficacy and safety of Cettum (Electric moxibustion) for patients with knee osteoarthritis.

DETAILED DESCRIPTION:
The investigator targets the patients with knee osteoarthritis. After treatment in 3 groups - Cettum treatment, traditional indirect moxibustion treatment, and usual care groups - the investigators will compare the effects of pain relieving and daily performing improvement. So the investigators will confirm the efficacy of Cettum, and further the best treatment method. In addition, the investigators are going to evaluate the safety of abnormal reaction during the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. At least 40 years of age, but below 70 years of age
2. Presence of knee osteoarthritis diagnosed according to American College of Rheumatology classification criteria and satisfying the following 2 conditions

   * Knee pain when weight load in one or both knees in the last 6 months

     * Knee pain rated >4cm on a 10cm Visual Analog Scale (VAS)
3. Feeling temperature sense to distinguish temperature differences
4. An understanding of the objectives and methods of the clinical trial, and willingness in completing the consent form
5. Those who are reliable and willing to cooperate in this test, and obey the restrictions for the next 3 months

Exclusion Criteria:

1. Trauma to the knee(s) within 6 months prior to enrollment, causing pain or functional problems
2. Surgery on the knee(s) within 6 months prior to enrollment, causing pain or functional problems
3. A history of intra-articular injection within the last 3 months
4. A physical or laboratory finding indicating presence of an inflammatory arthritis (e.g. rheumatoid arthritis, autoimmune disease)
5. Presence of physical or psychiatric disorder that may affect moxibustion treatment
6. Presence of neurological disorder including paralysis symptoms on local or general sensation
7. A female who is pregnant or is lactating
8. Being afraid of moxibustion treatment or expected to cause side effects
9. When researchers evaluate that it is not appropriate to participate in this clinical test

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Pain NRS (Numeric Rating Scale) change | 6 weeks
  The Numeric Rating Scale is a unidimensional measure of pain intensity. The 11-point numeric scale ranges from '0' representing 'no pain' to '10' representing 'worst pain imaginable'.

SECONDARY OUTCOMES:
100mm Pain VAS (Visual Analogue Scale) | 6 weeks
  The patient is asked to indicate their perceived pain intensity along a 100mm horizontal line, where '0' represents 'no pain' and '100', 'unbearable pain'.
WOMAC (Western Ontario and McMaster Universities) total | 6 weeks
  WOMAC scale is widely used to evaluate the condition of patients with osteoarthritis of the knee, including pain, stiffness, and physical functioning of the joints. The WOMAC scale measures 5 items for pain, 2 for stiffness, and 17 for functional limitation.
EQ-5D-5L (EuroQol 5-Dimensions 5-Levels) | 6 weeks
  The EQ-5D-5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
PGA (Patient Global Assessment) | 6 weeks
  The patient may choose to answer the question of how much better the symptom has improved compared to the previous treatment: Very good, Good, Fair, Poor, Very poor.
Temperature sense threshold | 6 weeks
  Investigator attaches the temperature sensor to the measurement area and increase or decrease the temperature by starting with reference temperature. Warm pain threshold and heat pain threshold are recorded to compare the difference between the value at baseline and the value at the end of the treatment.
Adverse Events | 6 weeks
  Any unpredicted symptoms are checked at each visit and if any, the symptom, time of occurrence, and length of duration are recorded and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Eun Jung Kim, Ph. D., Principal Investigator — DongGuk University
Locations (2):
- South Korea (2):
  - Dongguk University Ilsan Oriental Hospital, Goyang-si, Gyeonggi-do
  - Dongguk University Bundang Oriental Hospital, Seongnam-si, Gyeonggi-do

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang HR, Jung CY, Lee SD, Kim KH, Kim KS, Kim EJ. Efficacy and safety of electrical moxibustion for knee osteoarthritis: study protocol for a randomized controlled trial. Trials. 2018 Mar 5;19(1):159. doi: 10.1186/s13063-018-2514-x. PMID 29506572